CLINICAL TRIAL: NCT02470598
Title: PD-Improved Dialysis Efficiency With Adapted APD - PD-IDEA
Brief Title: PD-Improved Dialysis Efficiency With Adapted APD
Acronym: PD-IDEA
Status: Completed | Type: Observational
Sponsor: Fresenius Medical Care Deutschland GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: PD-aAPD-01-INT
Record Dates: First submitted 2015-04-28; First posted 2015-06-12 (Estimated); Last update posted 2020-08-06 (Actual); Status verified 2020-07

CONDITIONS: Chronic Renal Failure
Keywords: Automated Peritoneal Dialysis; Adapted APD (aAPD); Hydration status; Residual Renal Function; Ultrafiltration
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Therapeutics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Treatment with Adapted Automated Peritoneal Dialysis (aAPD) — This is a purely non-interventional, observational study, where treatment decisions are completely guided by the discretion of the attending nephrologists

SUMMARY:
The aim of this study is to observe the effect of adapted APD (aAPD) on maintenance and/or improvement of the hydration status of more than 250 PD patients, and to observe the tolerability of the therapy over a long period.

DETAILED DESCRIPTION:
In some studies it has been observed that the use of a combination of short dwell/small volume and long dwell/large volume can improve the effectiveness of APD. However, these studies have been performed in a small number of patients during a short observation period.

The aim of this study is to assess the hydration status of PD patients treated with aAPD and observe its development during one year using the BCM-Body Composition Monitor (BCM), a bioimpedance spectroscopy (BIS) device. In addition, it is intended to observe the variability of aAPD prescriptions and their influence on the hydration status of the patients.

This is a purely non-interventional, observational study, where treatment decisions are completely guided by the discretion of the attending nephrologists.

ELIGIBILITY:
Inclusion Criteria:

* CKD patients with indication for renal replacement therapy
* Patient treated or to be treated with aAPD
* Fluid status regularly monitored with BCM

Exclusion Criteria:

* Patients who have any condition prohibiting the use of BCM like patients with major amputations (e.g. lower leg)
* Participation in an interventional study which could have an effect on the study objectives hydration status and dialysis adequacy (e.g. studies on PD solutions, studies on diuretics)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic kidney disease (CKD) being treated or starting renal replacement therapy with aAPD
Sampling Method: Non-Probability Sample
Enrollment: 182 (Actual)
Dates: Start 2015-03; Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Hydration status | Every three months during one year
  Assessed via body composition measurements

SECONDARY OUTCOMES:
Residual renal function | Every three months during one year
Changes in prescription | Every three months during one year
Achievement of adequate solute removal | Every three months during one year
Therapy tolerability | Every three months during one year

OTHER OUTCOMES:
Change of therapy modality | Every three months during one year

CONTACTS AND LOCATIONS:
Overall Officials: Michel Fischbach, Prof., Study Director — University Hospital Hautepierre; Manel Vera, Dr., Study Director — Hospital Clinic i Provinvial de Barcelona; Emilio Galli, Dr., Study Director — Ospedale "Treviglio-Caravaggio" di Treviglio; Cecile Courivaud, Dr., Study Director — University Hospotal Besancon; Virpi Rauta, Dr., Study Director — Helsinki Univerity Hospital
Locations (50):
- Czechia (10):
  - Faculty Hospital Brno-Bohunice, Brno
  - Hospital Liberec, Liberec
  - Regional Hospital in Mlada Boleslav, Mladá Boleslav
  - Hospital Nove Mesto na Morave, Nové Město na Moravě
  - Faculty Hospital Pilsen, Pilsen
  - Faculty Hospital Karlovo namesti, Prague
  - Faculty Hospital Strahov, Prague
  - NC centre Vinohrady, Prague
  - NC centre Sokolov, Sokolov
  - Hospital Trebic, Třebíč
- Regional Hospital Viborg, Viborg, Denmark
- Finland (3):
  - Helsinki University Hospital, Helsinki
  - Kymenlaakso Central Hospital, Kotka
  - Regional Hospital Roskilde, Lappeenranta
- Malaysia (5):
  - Hospital Selayang, Batu Caves
  - Gleneagles Hospital Kuala Lumpur (GHKL), Kuala Lumpur
  - Hospital Universiti Kebangsaan Malaysia (HUKM), Kuala Lumpur
  - Hospital Serdang, Serdang
  - Hospital Seremban, Seremban
- Spain (24):
  - Complejo Hospitalario universitario de Albacete, Albacete
  - Fundación Hospital de Alcorcón, Alcorcón
  - Complejo Asistencial de Avila, Ávila
  - Fundacion Puigvert, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital de Basurto, Bilbao
  - Hospital General de Castellón, Castellon
  - Hospital Universitario di Girona Josep Trueta, Girona
  - Hospital General Virgen de las Nieves, Granada
  - Complejo hospitalario de Jaén, Jaén
  - Complejo Hospitalario San Millán-San Pedro De La Rioja, Logroño
  - Hospital Universitario Lucus Agusti, Lugo
  - Hospital Clínico San Carlos, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Universitario Puerta de Hierro, Majadahonda
  - Hospital Carlos Haya, Málaga
  - Complexo Hospitalario Universitario de Ourense (CHUO), Ourense
  - Hospital Universitario Central de Asturias (HUCA), Oviedo
  - Hospital Universitatio Donostia, San Sebastián
  - Complejo Hospital Universitario de Santiago (CHUS), Santiago de Compostela
  - Hospital Clínico de Valencia, Valencia
  - Hospital Peset, Valencia
  - Hospital Universitari i Politècnic La Fe, Valencia
  - Hospital Txagorritxu, Vitoria-Gasteiz
- Sweden (7):
  - Danderyds Sjukhus AB, Danderyd
  - Höglandssjukhuset Eksjö/Nässjö, Eksjö
  - Kalmar Hospital, Kalmar
  - Skåne University Hospital, Lund
  - Länssjukhuset Sundsvall, Sundsvall
  - Norra Älvsborgs Länssjukhus, Trollhättan
  - Norrlands University Hopsital, Umeå